CLINICAL TRIAL: NCT04302558
Title: Low-Intensity Blood Flow Restriction Training as a Pre-Operative Rehabilitative Modality to Improve Post-Operative Outcomes for ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Anikar Chhabra, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19-008473
Record Dates: First submitted 2020-03-08; First posted 2020-03-10 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction (BFR) group (Experimental): Subjects previously diagnosed with a torn ACL who have yet to undergo surgical reconstruction and pre-operative rehabilitation will do a series of low-intensity strength exercises while the blood flow to the leg is reduced by a blood flow restriction cuff.
  Interventions: Behavioral: Exercise Blood Flow Restriction training
- SHAM Blood Flow Restriction (BFR) group (Sham Comparator): Subjects previously diagnosed with a torn ACL who have yet to undergo surgical reconstruction and pre-operative rehabilitation will do a series of low-intensity strength exercises while a blood flow restriction cuff is applied but inflation pressure will be limited
  Interventions: Behavioral: SHAM Exercise Blood Flow Restriction training

INTERVENTIONS:
Behavioral: Exercise Blood Flow Restriction training — While exercising, an Inflatable cuff, similar to a blood pressure cuff, is applied to the proximal aspect of the femur of the affected lower extremity inflated to occlude blood flow
  Arms: Blood Flow Restriction (BFR) group
Behavioral: SHAM Exercise Blood Flow Restriction training — While exercising Inflatable cuff, similar to a blood pressure cuff, applied to the proximal aspect of the femur of the affected lower extremity with limited inflation pressure to not occlude blood flow
  Arms: SHAM Blood Flow Restriction (BFR) group

SUMMARY:
Researchers are trying to find out whether the use of low-intensity strength exercises during the 2 weeks before surgery, and while the blood flow to the leg is reduced, will improve the outcomes after surgery to repair an injured ligament of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between 13 and 40 years old
* Subjects must have been previously diagnosed with a tear of the anterior cruciate ligament in one of the lower extremities that requires surgical reconstruction
* Subjects must be able to understand study procedures and comply with them for the entire duration of the study
* Subjects must have normal contralateral limb strength

Exclusion Criteria:

* Subjects with any personal history of deep vein thrombosis or with such history in their immediate family
* Subjects who have any multi-ligamentous injuries to the knee that require modified post-operative unloading
* Subjects who have history of previous anterior cruciate ligament reconstructions in either the affected or unaffected leg
* Subjects with an inability or unwillingness of individual or legal guardian to give written informed consent

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Change in muscle diameter (hypertrophy) | 2 weeks pre-operative, 8-10 days post-operative
  Measured using ultrasound images of the musculature and soft tissue of the quadriceps femoris

SECONDARY OUTCOMES:
Change in muscle strength | 2 weeks pre-operative, 4 weeks pre-operative, 8 weeks post-operative
  Muscle strength will be measured in subjects as the percent strength of the injured leg compared to the non-injured leg based on handheld dynamometer and the number of leg presses performed at the 1-rep maximum

CONTACTS AND LOCATIONS:
Overall Officials: Anikar Chhabra, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGurren DP, Glattke KE, Chhabra A, Boddu SP, Poon SK, Flug JA, Brinkman JC, Goetzinger S, Lee JE, Nocella A, Rogge J, De Luigi AJ. Assessment of Interrater Reliability for Interpretation of Musculoskeletal Ultrasound Imaging of the Quadriceps Femoris. Am J Phys Med Rehabil. 2025 Oct 1;104(10):906-910. doi: 10.1097/PHM.0000000000002731. Epub 2025 Mar 6. PMID 40101801
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials